CLINICAL TRIAL: NCT05739552
Title: Telerehabilitation in the Post-COVID-19 Patient: the Italy-Switzerland Experience
Brief Title: Telerehabilitation in the Post-COVID-19 Patient (TRIALS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 31A101
Record Dates: First submitted 2023-02-20; First posted 2023-02-22 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation (Experimental)
  Interventions: Other: Telerehabilitation program

INTERVENTIONS:
Other: Telerehabilitation program — Application of customised respiratory and/or motor rehabilitation exercises to be carried out directly at the patients' home after hospital discharge in order to evaluate its effects.

SUMMARY:
A major issue brought about by the current pandemic concerns the discontinuation of a large proportion of outpatient services provided locally, especially in the rehabilitation field. Added to this situation is the ever-increasing demand for rehabilitation for post-COronaVIrus Disease 19 (COVID-19) patients. Data show that respiratory and motor rehabilitation for people infected with COVID-19 is necessary at all stages of the disease, even in the medium to long term after discharge from acute hospital care. Also to be taken into account are the logistical difficulties imposed by restrictions on the movement of individuals within the territory for both patients and caregivers, which are amplified in remote or poorly served areas, such as many cross-border territories. In this context, telerehabilitation can provide solutions to assist healthcare facilities in managing the demand for rehabilitation in the territory using a 'digital' therapist. The main objective of this project is therefore to identify the appropriate technology to administer the rehabilitation programme to patients and apply to a group of post-COVID-19 patients a customised respiratory and/or motor rehabilitation programme to be carried out directly at the patients' home after hospital discharge in order to evaluate its effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to a rehabilitation facility for functional recovery in disabling motor and/or respiratory outcomes of severe acute respiratory syndrome COronaVirus 2 (SARS-CoV2) infection and residing in cross-border regions with a low density of rehabilitation offerings.

Exclusion Criteria:

* Psychiatric disorders/cognitive impairments that do not allow proper use of tablets and breathing training devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline aerobic endurance. | up to 8 weeks
  Measurement of aerobic endurance using the six-minutes walk test (6MWT) at baseline (upon admission, T0), 3-4 weeks later after multidisciplinary rehabilitation + respiratory and motor training (at discharge, T1) and after 3-4 weeks of telerehabilitation (T2).
Change from baseline balance and functional mobility. | up to 8 weeks
  Measurement of balance and functional mobility using Timed Up and Go test (TUG) at baseline (upon admission, T0), 3-4 weeks later after multidisciplinary rehabilitation + respiratory and motor training (at discharge, T1) and after 3-4 weeks of telerehabilitation (T2).
Change from baseline isometric strength. | up to 8 weeks
  Measurement of isometric strength using the handgrip test (kg) at baseline (upon admission, T0), 3-4 weeks later after multidisciplinary rehabilitation + respiratory and motor training (at discharge, T1) and after 3-4 weeks of telerehabilitation (T2).
Change from baseline in several respiratory measures. | up to 8 weeks
  Performing force vital capacity (FVC), maximum inspiratory (MIP) and expiratory (MEP) pressure and two one-minute maximum voluntary ventilation respiratory tests with the SpiroTiger device (first test with a ventilatory rate of 26 acts/min with increased load on the inspiratory muscles and second test with a ventilatory rate of 34 acts/min with increased load on the expiratory muscles) at baseline (upon admission, T0), 3-4 weeks later after multidisciplinary rehabilitation + respiratory and motor training (at discharge, T1) and after 3-4 weeks of telerehabilitation (T2).
Change from baseline in the pulmonary function test. | up to 8 weeks
  Performing a spirometry test with diffusing capacity of the lungs for carbon monoxide (DLCO) at baseline (upon admission, T0), 3-4 weeks later after multidisciplinary rehabilitation + respiratory and motor training (at discharge, T1) and after 3-4 weeks of telerehabilitation (T2).

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Cimolin, Principal Investigator — Politecnico di Milano
Locations (2):
- Istituto Auxologico Italiano IRCCS, Oggebbio, VB, Italy
- Clinica Hildebrand, Brissago, Switzerland

IPD SHARING:
Plan to Share IPD: No